CLINICAL TRIAL: NCT01664624
Title: A Phase 1b, Randomized, Double-Blind, Active Comparator (Open-Label Exenatide) Controlled Study to Evaluate the Effect of Roflumilast Plus Alogliptin on Postprandial Active GLP-1 Level and 24-hour Glucose Level in Subjects With Type 2 Diabetes Who Are Inadequately Controlled on a Stable Dose of Metformin
Brief Title: Roflumilast Plus Alogliptin Proof-of-Mechanism Study in Type2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-T2D_107; U1111-1128-6945 (Registry Identifier: WHO)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Roflumilast; alogliptin; Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Roflumilast + alogliptin (Experimental): Roflumilast 500 μg, tablets, orally and alogliptin 25 mg, tablets, orally, once a day for 11 days.
  Interventions: Drug: Roflumilast; Drug: Alogliptin
- Alogliptin alone (Experimental): Placebo to roflumilast, tablets, orally and alogliptin, 25 mg, tablets, orally, once a day for 11 days.
  Interventions: Drug: Alogliptin; Drug: Placebo to roflumilast
- Roflumilast alone (Experimental): Roflumilast 500 μg, tablets, orally and placebo to alogliptin, tablets, orally, once a day, for 11 days.
  Interventions: Drug: Roflumilast; Drug: Placebo to alogliptin
- Exenatide (Active Comparator): Exenatide 5 μg subcutaneous injection twice a day for 11 days.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Roflumilast — Roflumilast tablets
  Other Names: Daxas, Daliresp
  Arms: Roflumilast + alogliptin; Roflumilast alone
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina
  Arms: Alogliptin alone; Roflumilast + alogliptin
Drug: Exenatide — Exenatide solution
  Other Names: Byetta; Bydureon
  Arms: Exenatide
Drug: Placebo to roflumilast — Placebo-matching roflumilast tablets
  Arms: Alogliptin alone
Drug: Placebo to alogliptin — Placebo-matching alogliptin tablets
  Arms: Roflumilast alone

SUMMARY:
The purpose of this study is to assess the effect of roflumilast plus alogliptin on glucagon-like peptide-1 (GLP-1) and glucose levels in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This is a study to evaluate the antiglycemic efficacy and safety of roflumilast + alogliptin compared to alogliptin alone and roflumilast alone; it will also include an open-label exenatide treatment arm as a control. The antiglycemic efficacy of the combination will be evaluated through the measurement of postprandial active GLP-1 level, ß cell secretion activity (via the measurement of C-peptide and insulin levels), appetite sensations (as assessed by VAS) and glycemic control as assessed by a continuous glucose monitoring system (CGMS).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 80 years, inclusive, at the time of dosing on Day 1.
2. Has an historical diagnosis of type 2 diabetes mellitus (T2DM) disease.
3. Has a documented history of a diet and exercise plan and is receiving metformin as monotherapy at a stable dose for at least 8 weeks prior to Screening; has no chronic use (>7 days) of any other antidiabetic therapy within the 8 weeks prior to Screening.
4. Has inadequate glycemic control at Screening, as evidenced by HbA1c (glycosylated hemoglobin) level between 7.0% and 10.0%, inclusive.
5. Has a body mass index (BMI) of ≥23.0 kg/m^2 and ≤45.0 kg/m^2, at Screening.
6. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
7. A male who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose of study drug
8. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
9. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Has a history of type 1 diabetes.
2. Has a history of acute metabolic diabetic complications.
3. Has has abnormal Screening or Check-in (Day -2) laboratory values that suggest a clinically significant underlying disease (eg, active liver disease or jaundice) or participant with the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN).
4. Has a history of diabetic gastroparesis or history of gastric bypass surgery.
5. Has a history of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months prior to Screening.
6. Has New York Heart Association heart failure of Class (III-IV) regardless of therapy.
7. Has a supine blood pressure >150 mm Hg for systolic or >90 mm Hg for diastolic, confirmed on repeat testing within a maximum of 5 minutes, at Screening and Check-in (Day -2).
8. Has presence or history of neuropsychiatric disorder (eg, psychosis, psychotic disorders, depression associated with suicidal thinking, suicidal ideation or behavior).
9. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. Has a hemoglobin ≤120 g/L for men and ≤100 g/L for women.
11. Has a history of clinically significant allergies or idiosyncrasies to roflumilast, alogliptin and exenatide or any inactive ingredient(s) of these products, eg, rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, glucose-galactose malabsorption or phenylketonuria.
12. Has received alogliptin or roflumilast in a previous clinical study or as a therapeutic agent within 2 months prior to Screening, or is taking prescription roflumilast for chronic obstructive pulmonary disease (COPD), or has received any other investigational compound within 30 days prior to the first dose of study medication, or is participating or plans to participate in any other clinical trial during this study.
13. If female, is pregnant or lactating or intending to become pregnant before, during, or within 30 days after last dose; or intending to donate ova during such time period.
14. If male, intends to donate sperm during the course of the study or for 30 days after last dose of study medication.
15. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
16. Has a history of cancer, except basal cell or squamous cell carcinoma which has been in remission for at least 5 years prior to Day 1.
17. Serum creatinine ≥1.5 mg/dL for males and ≥1.4 mg/dL for females or creatinine clearance <60 mL/minutes, based on calculation by central lab using the Cockcroft-Gault approximation at Screening Visit.
18. Has a history of any hemoglobinopathy that may affect determination of HbA1c.
19. Has positive test result for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV), any known history of infection with human immunodeficiency virus (HIV), any acute infection, or severe immunological diseases (eg, multiple sclerosis, systemic lupus erythematosus, and progressive multifocal leukoencephalopathy).
20. Has a risk of suicide according to the Investigator's clinical judgment per Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or has made a suicide attempt in the past 6 months.
21. Has any clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation (as assessed by the investigator).
22. Does not have an adequate standard of literacy to allow him or her to complete the study diary during non-clinic days.
23. Has poor peripheral venous access.
24. Has Screening or Check-in (Day -2) abnormal clinically significant electrocardiogram (ECG). Entry of any participant with abnormal not clinically significant ECG must be approved and documented by signature of Principal Investigator and Medical Monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Chula Vista, California
  - Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 10 July 2012 to 29 November 2012.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus and inadequate glycemic control were enrolled equally in 1 of 4 treatment groups, roflumilast + alogliptin, alogliptin alone, roflumilast alone, or exenatide.
Period: Overall Study
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Started | 10 | 11 | 10 | 9
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide | Total
Number analyzed (Participants) | 10 | 11 | 10 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.15) | 52.9 (7.52) | 60.7 (4.24) | 54.6 (6.88) | 54.7 (8.15)
Age, Customized [Number; unit: participants]
  < 65 years | 10 | 11 | 9 | 9 | 39
  ≥ 65 years | 0 | 0 | 1 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 4 | 15
  Male | 6 | 8 | 6 | 5 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 7 | 6 | 7 | 6 | 26
  Non-Hispanic or Latino | 3 | 5 | 3 | 3 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 3 | 2 | 0 | 8
  White | 7 | 8 | 8 | 9 | 32
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 10 | 9 | 40
Height [Mean (Standard Deviation); unit: cm] | 171.1 (8.91) | 171.2 (6.03) | 166.6 (10.44) | 166.4 (5.90) | 169.0 (8.09)
Weight [Mean (Standard Deviation); unit: kg] | 103.12 (21.688) | 93.24 (11.670) | 89.33 (17.961) | 86.98 (14.713) | 93.32 (17.329)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.93 (4.708) | 31.75 (3.184) | 32.03 (5.311) | 31.37 (4.653) | 32.53 (4.548)
Smoking Classification [Number; unit: participants]
  Never smoked | 6 | 6 | 10 | 7 | 29
  Current smoker | 1 | 0 | 0 | 0 | 1
  Ex-smoker | 3 | 5 | 0 | 2 | 10
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.9 (4.63) | 8.5 (6.39) | 7.0 (3.86) | 8.2 (6.63) | 7.7 (5.33)
Metformin Dose [Mean (Standard Deviation); unit: mg] | 875.0 (151.38) | 745.0 (225.40) | 805.0 (220.42) | 855.6 (211.31) | 819.2 (202.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Postprandial Area Under the Curve From Time 0 to 8 Hours (AUC[0-8]) for Active Glucagon-like Peptide-1
Description: The concentration of glucagon-like peptide-1 (GLP-1) in blood before and up to 8 hours after eating (postprandial) was plotted and the area under the curve calculated using the linear trapezoidal rule at Baseline and on Day 11. Least squares means of the change from Baseline to Day 11 were obtained using an analysis of covariance (ANCOVA) model with treatment as fixed effect, and Baseline postprandial AUC (0-8) of active GLP-1 as a continuous covariate.
Time Frame: Baseline and Day 11; samples were taken at -15 min and -5 min (pre-meal), and 15 min, 30 min, and 1, 2, 3, 4, 6, and 8 hours (post-meal).
Population: Full analysis set defined as all randomized participants included in the safety analysis. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: pmol/L*hr
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
pmol/L*hr | 26.5 (4.04) | 31.6 (4.01) | 3.8 (3.94) | -2.3 (4.14)
Statistical Analysis 1: Comparison: Roflumilast + Alogliptin vs Alogliptin Alone; ANCOVA was used to test the null hypothesis that the change from Baseline in the postprandial AUC(0-8) of active GLP-1 is no difference between the roflumilast + alogliptin and alogliptin alone; Test type: Superiority or Other; p = 0.388, ANCOVA — The comparison was evaluated at the 5% level of significance; ANCOVA model with treatment as fixed effect, and baseline Postprandial AUC (0-8) of active GLP-1 as a continuous covariate; LS Mean Difference = -5.1, 95% CI 2-sided [-16.9 to 6.7], Standard Error of Mean 5.82
Statistical Analysis 2: Comparison: Roflumilast + Alogliptin vs Roflumilast Alone; ANCOVA was used to test the null hypothesis that the change from Baseline in the postprandial AUC(0-8) of active GLP-1 is no difference between the roflumilast + alogliptin and roflumilast alone; Test type: Superiority or Other; p < 0.001, ANCOVA — The comparison was evaluated at the 5% level of significance; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 22.7, 95% CI 2-sided [11.1 to 34.3], Standard Error of Mean 5.70
Statistical Analysis 3: Comparison: Roflumilast + Alogliptin vs Exenatide; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — The comparison was evaluated at the 5% level of significance; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 28.8, 95% CI 2-sided [17.1 to 40.5], Standard Error of Mean 5.76

2. Secondary Outcome: Change From Baseline in AUC(0-8) of Postprandial Plasma Glucose
Description: The concentration of glucose in blood before and up to 8 hours after eating (postprandial) was plotted and the area under the curve calculated using the linear trapezoidal rule at Baseline and on Day 11. Least squares means of the change from Baseline to Day 11 were obtained using an ANCOVA model with treatment as fixed effect, and baseline postprandial AUC (0-8) of plasma glucose as a continuous covariate.
Time Frame: Baseline and Day 11 at -15 min and -5 min (pre-meal), and 15 min, 30 min, and 1, 2, 3, 4, 6, and 8 hours (post-meal).
Population: Full analysis set. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: mmol/L*hr
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
mmol/L*hr | -13.4 (2.70) | -9.8 (2.71) | -9.0 (2.71) | -18.5 (2.85)

3. Secondary Outcome: Change From Baseline in Postprandial AUC(0-8) of C-peptide
Description: The concentration of C-peptide in blood before and up to 8 hours after eating (postprandial) was plotted and the area under the curve calculated using the linear trapezoidal rule at Baseline and on Day 11. Least squares means of the change from Baseline to Day 11 were obtained using an ANCOVA model with treatment as fixed effect, and Baseline postprandial AUC (0-8) of C-peptide as a continuous covariate.
Time Frame: as for outcome 1
Population: Full analysis set. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: ng/mL*hr
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
ng/mL*hr | 1.0 (1.15) | 1.4 (1.16) | -0.7 (1.17) | 0.0 (1.22)

4. Secondary Outcome: Change From Baseline in Postprandial AUC(0-8) of Insulin
Description: The concentration of insulin in blood before and up to 8 hours after eating was plotted and the area under the curve calculated using the linear trapezoidal rule at Baseline and on Day 11. Least squares means of the change from Baseline to Day 11 were obtained using an ANCOVA model with treatment as fixed effect, and Baseline postprandial AUC (0-8) of insulin as a continuous covariate.
Time Frame: as for outcome 1
Population: Full analysis set. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: pmol/L*hr
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
pmol/L*hr | -49.5 (181.09) | 107.8 (180.75) | 26.9 (180.38) | -136.4 (190.12)

5. Secondary Outcome: Change From Baseline to Day 11 in AUC(0-8) of Appetite Sensation
Description: Appetite sensations were measured using a visual analog scale (VAS) questionnaire. Participants were asked to indicate their level of fullness, hunger, satiety, and prospective consumption (how much do you think you can eat?) on a 100 mm line ranging from "Not at all" (0 mm) to "extremely" (100 mm). Appetite sensation scores before and up to 8 hours after eating were plotted and the area under the curve calculated using the linear trapezoidal rule at Baseline and on Day 11. Least squares means of the change from Baseline to Day 11 were obtained using an ANCOVA model with treatment as fixed effect, and Baseline postprandial AUC (0-8) of appetite sensation VAS score as a continuous covariate.
Time Frame: At Baseline and Day 11, every 30 minutes, starting 1 hour before eating until 8 hour after the meal.
Population: Full analysis set. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: mm*hr
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
mm*hr
  Fullness | 70.5 (59.73) | 62.0 (56.52) | 136.0 (57.81) | 116.8 (59.51)
  Hunger | -103.6 (52.61) | 3.1 (52.18) | -132.7 (52.44) | -122.5 (54.92)
  Prospective consumption | -97.1 (54.24) | -14.9 (53.76) | -169.5 (53.98) | -124.3 (56.53)
  Satiety | -82.7 (53.66) | -3.2 (52.96) | -139.2 (53.58) | -127.7 (55.80)

6. Secondary Outcome: Change From Baseline to Day 11 in 24-hour Average Plasma Glucose
Description: Plasma glucose was measured by Continuous Glucose Monitoring System (CGMS). CGMS measures glucose every 5 minutes, starting in the fasting state 8 hour prior to the standardized breakfast (12 AM) until 16 hours after the breakfast. The average 24-hour plasma glucose concentration was calculated. Least squares means were obtained using an ANCOVA model with treatment as fixed effect, and Baseline 24-hour Glucose Measured by CGMS as a continuous covariate.
Time Frame: Baseline (Day -1) and Day 11, from 12 AM through 24 hours.
Population: Full analysis set. Only participants with data at both Baseline and post-baseline visits are included.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Number analyzed (Participants) | 10 | 10 | 10 | 9
mg/dL | -25.4 (6.67) | -17.5 (6.67) | -14.5 (6.66) | -34.9 (7.02)

ADVERSE EVENTS:
Time Frame: From the first dose of study medication to no more than 30 days after the last dose of the study medication (a maximum of 41 days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Roflumilast + Alogliptin | Alogliptin Alone | Roflumilast Alone | Exenatide
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 6/10 | 5/11 | 8/10 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast + Alogliptin (N=10) | Alogliptin Alone (N=11) | Roflumilast Alone (N=10) | Exenatide (N=9)
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast + Alogliptin (N=10) | Alogliptin Alone (N=11) | Roflumilast Alone (N=10) | Exenatide (N=9)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 4 | 4
Nausea (Gastrointestinal disorders) | 2 | 1 | 5 | 2
Headache (Nervous system disorders) | 3 | 2 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.